CLINICAL TRIAL: NCT02749864
Title: Personalized Medicine in HCV Infection. A Prospective, Multicenter, Epidemiological Study to Evaluate the Prevalence of Hepatitis C Infection in Spain in 2015 (PREVHEP)
Brief Title: Study to Evaluate the Prevalence of Hepatitis C in Spain in 2015 (PREVHEP)
Acronym: PREVHEP
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: JCG-PREVHEP-2015-01
Record Dates: First submitted 2016-04-16; First posted 2016-04-25 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C; Hepatitis B
Keywords: Hepatitis; Prevalence; Epidemiology; Infectious diseases
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Hepatitis; Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of whole blood, plasma and serum will be collected to analyse different markers related to the virus and the medical status of the patients.
  DNA samples will be transferred to the Biobank Valdecilla (Node DNA and fluids) according to Spanish law. Law 14/2007 of 3 July, on biomedical research and the Biobank law:
  Royal Decree 1716/2011, establishing the basic requirements for authorization and operation of biobanks are established for biomedical research and treatment of biological samples of human origin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Age 20-34 yr: No intervention Cohort of subjects aged 20-34 years old.
- B: Age 35-49 yr: No intervention Cohort of subjects aged 35-49 years old.
- C: Age 50-79 yr: No intervention Cohort of subjects aged 50-79 years old.

SUMMARY:
The hypothesis of this investigation stresses that the current understanding of the prevalence of HCV infection in the general population and in different subgroups will serve to lay out medium- and long-term measures for action geared toward reducing the disease burden through preventive, research, screening and therapeutic measures.

Aim: To determine the prevalence of seropositivity and chronic infection with the HCV and to analyze the associated factors. To analyze and infer different screening strategies for HCV infection based on the at-risk groups/cohorts of elevated prevalence detected. to assess the efficiency of screening strategies and the subsequent cost-effectiveness of treatment in the general population

DETAILED DESCRIPTION:
Design of the study: Seroepidemiological and virological study of cross-sectional population-based.

Patients and sampling: The study population has been distributed in groups according to age (20-34; 35-49; 50-74 years) and sex. In order to select a representative sample of this overall population, three Spanish regions will be selected on the basis of their different HCV-related hospitalisation rates defined as follows: high, >120 cases/100,000 inhabitants (Madrid); medium, 90-119 cases/100,000 inhabitants (Cantabria); or low, <90 cases/100,000 inhabitants (Valencia).

The participants will be selected through a random, representative sample using our two-stage conglomerate sampling with stratification of the First-Stage Units. These FSUs are made up by the Basic Health Areas (Health Centers). The Second-Stage Units are made up by the individuals. The stratification criteria used in the first stage will be the socioeconomic status-rural/urban environment. The selection of sample elements will be carried out through simple random sampling from the healthcare card database pertaining to the selected Health Centers. A sequence of random, computer-generated numbers will be obtained.

Sample size: In order to achieve an accuracy of 0.4% in the estimate of a percentage through a two-tailed 95% confidence interval, assuming the prevalences indicated by age strata in the general Spanish population (0.6%, 1.9% and 2.7% respectively), a total of 12,263 subjects distributed as follows: 1,456 aged 20-34 years, 4,476 aged 35-49 years and 6,331 aged 50-74 years.

Anticipating an uptake of 9-15%,21 following invitation via telephone, between 81,753 and 136,255 subjects distributed over the three regions needed to be contacted at random.

Recruitment method for randomized patients. Selected subjects will be called by phone by trained personnel. The subject will be invited to report for an interview in order to carry out a socio-healthcare questionnaire, a physical examination, and an analytical test. In the event the patient refuses to participate, permission shall be requested to collect minimum anonymous data for the subsequent study of possible screening biases. Patients meeting inclusion criteria and provide written informed consent to be included in the study.

Variables in the study: socio-healthcare questionnaire includes variables such as age, sex, socioeconomic status, risk factors, health habits, etc. Analytical variables (blood count, biochemistry, serologies for HBV and HCV, etc.) are collected. A Fibroscan is also performed. A cost-effectiveness of screening strategies and treatment will be analysed using a Markov model

Full duration: 21 months

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 74 who have health card in each of the autonomous communities studied.
* They agree to participate, understand and give informed consent.

Exclusion Criteria:

* Do not meet the criteria above.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population aged 20-74 years who agree to participate when contacted by phone call after a two-stage conglomerate sampling with stratification of the First-Stage Units.
  The study will be carried out in three Autonomous Communities (regions) in Spain.
Sampling Method: Probability Sample
Enrollment: 12246 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Serum Anti-HCV | 1 day
  Anti-HCV seroprevalence

SECONDARY OUTCOMES:
HCV RNA viral load | 1 day
  Chronic HCV infection
Serum HBsAg | 1 day
  HBV portador status
Birth date | 1 day
  Questionnaire about socio-economic and Health variables
Sex | 1 day
  Questionnaire about socio-economic and Health variables
Nationality | 1 day
  Questionnaire about socio-economic and Health variables
Residence time in Spain | 1 day
  Questionnaire about socio-economic and Health variables
Educational level | 1 day
  Questionnaire about socio-economic and Health variables
Activity and professional qualifications | 1 day
  Questionnaire about socio-economic and Health variables
Lifestyle habit/risk factor score | 1 day
  Questionnaire about socio-economic and Health variables
Nosocomial risk score | 1 day
  Questionnaire about socio-economic and Health variables
History of previous check of HCV/HBV exposure | 1 day
  Questionnaire about socio-economic and Health variables
Sexual behaviour | 1 day
  Questionnarie about socio-economic and Health variables
Number of sexual partners | 1 day
  Questionnaire about socio-economic and Health variables
Weight (kg) | 1 day
  Weight (Anthropometric variables)
Height (cm) | 1 day
  Height (Anthropometric variables)
BMI | 1 day
  Body Mass Index (Anthropometric variables)
Abdominal perimeter (cm) | 1 day
  Abdominal perimeter (Anthropometric variables)
Waist perimeter (cm) | 1 day
  Waist perimeter (Anthropometric variables)
Blood pressure (mmHg) | 1 day
  Blood pressure
ALT | 1 day
  Liver function tests
AST | 1 day
  Liver function tests
Alkaline Phosphatase (AP) | 1 day
  Liver function tests
GGT (Gammaglutamyl transferase) | 1 day
  Liver function tests
Bilirubin | 1 day
  Liver function tests
Serum Albumin | 1 day
  Biochemistry parameters
Total Cholesterol | 1 day
  Biochemistry parameters
LDL Cholesterol | 1 day
  Biochemistry parameters
HDL Cholesterol | 1 day
  Biochemistry parameters
Triglycerides | 1 day
  Biochemistry parameters
White blood cell count (WBC or leukocyte count) | 1 day
  CBC
Hemoglobin | 1 day
  CBC
Platelets | 1 day
  CBC
INR | 1 day
  International Normalized Ratio
kPa in Fibroscan | 1 day
  Liver stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crespo García, MDPhD, Study Director — Head of Gastroenterology and Hepatology at Hospital Universitario Marqués de Valdecilla. Professor at the Universidad de Cantabria; Jose L Calleja, MDPhD, Principal Investigator — Head of Gastroenterology and Hepatology at Hospital Universitario Puerta de Hierro-Majadahonda; Miguel A Serra, MDPhD, Principal Investigator — Gastroenterology and Hepatology Department at Hospital Clínico U. de Valencia
Locations (3):
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Puerta de Hierro-Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruguera M, Forns X. [Hepatitis C in Spain]. Med Clin (Barc). 2006 Jun 17;127(3):113-7. doi: 10.1157/13090276. Spanish. PMID 16828003
- [Background] Ditah I, Ditah F, Devaki P, Ewelukwa O, Ditah C, Njei B, Luma HN, Charlton M. The changing epidemiology of hepatitis C virus infection in the United States: National Health and Nutrition Examination Survey 2001 through 2010. J Hepatol. 2014 Apr;60(4):691-8. doi: 10.1016/j.jhep.2013.11.014. Epub 2013 Nov 27. PMID 24291324
- [Background] McGarry LJ, Pawar VS, Panchmatia HR, Rubin JL, Davis GL, Younossi ZM, Capretta JC, O'Grady MJ, Weinstein MC. Economic model of a birth cohort screening program for hepatitis C virus. Hepatology. 2012 May;55(5):1344-55. doi: 10.1002/hep.25510. Epub 2012 Mar 18. PMID 22135116
- [Derived] Ezcurra I, Puente A, Cuadrado A, Tamayo I, Iruzubieta P, Arias-Loste MT, Gonzalez FJ, Pellon R, Sanchez S, Crespo J, Acebo M, Lopez-Hoyos M, Perez R, Cuesta A, Anton A, Echavarria V, Fabrega E, Crespo J, Fortea JI. No evidence of association between inherited thrombophilia and increased risk of liver fibrosis. United European Gastroenterol J. 2023 Dec;11(10):1010-1020. doi: 10.1002/ueg2.12500. Epub 2023 Nov 28. PMID 38015591
- [Derived] Llop E, Iruzubieta P, Perello C, Fernandez Carrillo C, Cabezas J, Escudero MD, Gonzalez M, Hernandez Conde M, Puchades L, Arias-Loste MT, Serra MA, Crespo J, Calleja JL. High liver stiffness values by transient elastography related to metabolic syndrome and harmful alcohol use in a large Spanish cohort. United European Gastroenterol J. 2021 Oct;9(8):892-902. doi: 10.1002/ueg2.12109. Epub 2021 Jun 2. PMID 34077628